CLINICAL TRIAL: NCT03451006
Title: (MATE) Metformin and Aging Trial in the Elderly: A Pilot and Feasibility Study
Brief Title: Effect of Metformin on Frailty in 12 Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficult recruitment and not achieved
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mandeep Singh, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-003088
Record Dates: First submitted 2018-01-30; First posted 2018-03-01 (Actual); Results first posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-10

CONDITIONS: Aging; Inflammation; Frailty
MeSH Terms: conditions — Inflammation; Frailty | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Arms Assigned interventions Placebo Comparator: Metformin Chronic metformin administration through augmentation of cellular regeneration and reduction of senescence will improve frailty and physical functioning as studied by the short physical performance battery (SPPB) test. Drug: Metformin versus placebo This will be a pilot, feasibility study. Twelve subjects ≥60 years with stable CAD and prediabetes, who score <9 on SPPB test will be randomized to receive up to 2gm of oral metformin or placebo for 12 months.
  Placebo comparator: Placebo Placebo will be compared to chronic metformin administration Drug: Metformin versus placebo This will be a pilot, feasibility study. Twelve subjects ≥60 years with stable CAD and prediabetes, who score <9 on SPPB test will be randomized to receive up to 2gm of oral metformin or placebo for 12 months.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Metformin 500mg tablet by mouth, every 6 to 8 hours for one year
  Interventions: Drug: Metformin
- Placebo (Active Comparator): Placebo by mouth every 6 to 8 hours for one year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Oral metformin (up to 2gm) will be given in divided doses
  Arms: Metformin
Drug: Placebo — Oral Placebo will be given in divided doses
  Arms: Placebo

SUMMARY:
This study will test whether chronic metformin administration will improve longevity of the cell, improves its machinery by reducing aging-related biochemical parameters and thereby improving physical performance, as measured by short physical performance battery test.

DETAILED DESCRIPTION:
Heart disease is the number one cause of death in the United States and disproportionately affects older adults, underscoring the need to examine determinants of survivorship. Recognizing this gap, current guidelines lay emphasis to assess frailty, a key construct prevalent in elderly and known to impact their prognosis.Older persons are commonly frail, manifest hyperglycemia and their health span is truncated by illnesses during which physiological declines together with accumulation of additional deficits results in multimorbidity and functional dependence. High incidence of functional decline and stress hyperglycemia in patients with coronary artery disease (CAD) makes pharmacologic manipulation, an attractive strategy to improve frailty and reduce adverse cardiovascular outcomes. Metformin exerts its effect on health span as a calorie restriction-mimetic through inhibition of mitochondrial complex 1 and activation of activated protein kinase (AMP).This drug is safe and has been shown to prolong life in mammals. Metformin by reducing effects of cellular senescence and improving glycemic control may improve the functioning of older adults.

In CAD, cellular senescence and inflammation affect organ dysfunction through interference with tissue homeostasis and regeneration. The deleterious effect of senescence includes pro-inflammatory senescence-associated secretory phenotype (SASP). Normal biological function through alteration in cellular homeostasis and restoration of glycemic control may be achieved by metformin. The phenotypic manifestations of these changes are incompletely characterized as it is yet unknown whether cell-intrinsic regenerative mechanisms can be translated into clinical improvement in physical performance and whether it's chronic administration is safe in older adults. These major gaps in knowledge hinder utilization of metformin as an agent to promote cellular regeneration and to reduce the impact of cellular senescence.

Targeting frail individuals with high levels of inflammation and SASP factors would necessitate identification of predictors of improvement with metformin in tissue inflammation and function. A clinomics approach implementing simultaneous assessment of clinical impact coupled with serological profiling would provide enhanced understanding of the local and systemic impact mediated by metformin. Through correlation of molecular profiles with phenotypic expression changes, as proposed herein, investigators will enhance understanding of the regenerative impact of metformin and the basis for clinical improvement in the setting of senescence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Stable CAD
* Prediabetes (one of the following criteria should be met)

  * Fasting plasma glucose: 100-126 mg/dL
  * HbA1C: 5.7-6.4
* Frailty (Short Physical Performance Battery: Score <9)
* Able to return for follow-up
* Written informed consent

Exclusion criteria:

* Pre-existing or new-onset diabetes
* Any active malignancy, hematological disorder, post organ transplant, immunocompromised
* Cancer requiring treatment in the past 3 years (other than non-melanoma skin cancer)
* Dementia [mini mental state examination (MMSE <20)]
* Disability (need for assistance in >2 of any six activities on Katz activities of daily living (ADL)46
* Prior stroke with disability
* Acute coronary syndrome <3months or participating in cardiac rehabilitation
* Severe Parkinson's
* Hepatic insufficiency and/or chronic liver disease (cirrhosis)
* Chronic kidney disease (GFR < 45 mL/min)
* Taking metformin for any indication
* Acute alcohol intoxication
* Known hypersensitivity to metformin hydrochloride
* Acute/chronic metabolic acidosis, including diabetic ketoacidosis, with or without coma

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Singh, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No plan to do that

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Metformin 500mg tablet by mouth, every 6 to 8 hours for one year
  Metformin: Oral metformin (up to 2gm) were given in divided doses
- Placebo: Placebo by mouth every 6 to 8 hours for one year
  Placebo: Oral Placebo were given in divided doses
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 4 | 3
Completed | 2 | 1
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Full Range); unit: years] | 75.75 [64.0 to 86.0] | 77.33 [71.0 to 81.0] | 76.54 [64.0 to 86.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Frailty
Description: Frailty will be measured by the Short Physical Performance Battery (SPPB). The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). Frailty is defined as a score of <9.
Time Frame: Baseline, 12 months
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Balance Score Standing With Feet Close Together
Description: This measure is part of the SPPB. The scores range from 0 (not attempted), to 2 (held for 10 seconds). Ability to stand longer in this position indicates greater balance.
Time Frame: Baseline, 12 months
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Balance Score Standing in Semi Tandem Position
Description: This measure is part of the SPPB. The semi tandem position is the heel of one foot place by the big toe of the other foot. The scores range from 0 (not attempted), to 2 (held for 10 seconds). Ability to stand longer in this position indicates greater balance.
Time Frame: Baseline, 12 months
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change in Balance Score Standing in Full Tandem Position
Description: This measure is part of the SPPB. The full tandem position is with the feet directly in front of each other. The scores range from 0 (not attempted), to 2 (held for 10 seconds). Ability to stand longer in this position indicates greater balance.
Time Frame: Baseline, 12 months
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Change in Gait Speed
Description: This measure is part of the SPPB. Subjects will be asked to walk 8 feet or 2.44 meters at their usual pace. They will be allowed to use a cane or other walking aid if it is their custom. Scores range from 0 = could not do to 4 =<3.1 seconds.
Time Frame: Baseline, 12 months
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Change in Score, Standing Test From Chair
Description: This measure is part of the SPPB. Subjects will be asked to try to stand up from a chair 5 times with arms folded across their chest, and will be timed. Scores range from 0 to 4, with 0 = unable to stand without using arms, and 4 = completing 5 stands in <11.1 seconds.
Time Frame: Baseline,12 months
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Interleukin 6 (pg/ml)
Description: Serum will be collected to measure the effect of metformin on senescent markers.
Time Frame: Baseline, 12 months
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Matrix Metalloproteinase (ng/ml)
Description: Serum will be collected to measure the effect of metformin on senescent markers.
Time Frame: Baseline, 12 months
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Plasminogen Activator Inhibitor
Description: Serum will be collected to measure the effect of metformin on senescent markers.
Time Frame: Baseline, 12 months
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Monocyte Chemotactic Protein-1
Description: Serum will be collected to measure the effect of metformin on senescent markers.
Time Frame: Baseline, 12 months
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in Activin
Description: Serum will be collected to measure the effect of metformin on senescent markers.
Time Frame: Baseline, 12 months
Population: Study was terminated due to recruitment being difficult and not achieved. Data was not collected nor analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 12 weeks
Description: Study was terminated due to recruitment being difficult and not achieved.
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

LIMITATIONS AND CAVEATS:
Study was terminated due to recruitment being difficult and not achieved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT03451006/Prot_000.pdf